CLINICAL TRIAL: NCT06843538
Title: Peri-operative Tamsulosin and Impact on Voiding Trial Following Outpatient Urogynecology Surgery: a Randomized Controlled Trial
Brief Title: Peri-operative Tamsulosin and Impact on Voiding Trial After Same-day Urogynecology Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 24-108
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Urinary Retention (POUR)
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Arm (Active Comparator)
  Interventions: Drug: Tamsulosin
- Control Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — This intervention will investigate if tamsulosin will decrease postoperative urinary retention. Subjects will be directed to start taking the medication 5-7 days prior to their procedure; as previous studies have shown, this is when tamsulosin reaches its steady state. Patients will continue to take their assigned pills for 7 days postoperatively.
  Other Names: Flomax
  Arms: Study Arm
Drug: Placebo — This intervention will ensure blinding and an accurate measure of the real effect of tamsulosin.
  Arms: Control Arm

SUMMARY:
The purpose of this research study is to determine if taking tamsulosin preoperatively decreases your chances of being discharged after surgery with a Foley catheter (flexible tube that drains urine from the bladder into a collection bag).

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing any pelvic organ prolapse repair or incontinence surgery

Exclusion Criteria:

* Any surgery involving a non-urogynecologist
* Patients already on an alpha blocker
* Baseline hypotension
* History of syncope
* Postural orthostatic tachycardia syndrome (POTS)
* Non-English speaker or interpreter unavailable for Spanish-speaking patient
* Impaired cognition impeding proper consenting
* Any other medical contraindication for tamsulosin use
* History of urinary retention requiring continuous or intermittent catheterization
* Patients consented for the study but then due to intraoperative complication, routine voiding trial no longer indicated due to requiring indwelling catheter or intermittent catheterization on discharge will be excluded from primary outcome analysis
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Voiding trial on postoperative day 0 | Day of surgery
  Whether or not patients pass or fail their postoperative voiding trial

SECONDARY OUTCOMES:
Secondary postoperative urinary retention | 2 weeks following surgery
  Patients who develop urinary retention after discharge
Postoperative urinary tract infection | 30 days after surgery
  Patients who develop a urinary tract infection after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- TriHealth, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No